CLINICAL TRIAL: NCT04677530
Title: A Double-blind, Placebo-controlled, Randomized, Single Ascending Dose and Multiple Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ-40411813 in Healthy Japanese Adult Male Subjects
Brief Title: A Study of JNJ-40411813 in Healthy Japanese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108942; 40411813EDI1011 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2020-12-18; First posted 2020-12-21 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — 1-butyl-3-chloro-4-(4-phenyl-1-piperidinyl)-(1H)-pyridone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: JNJ-40411813 or Matching Placebo (Experimental): Participants will receive a single oral dose of JNJ-40411813 or a matching placebo in Cohorts 1, 2, and 3.
  Interventions: Drug: JNJ-40411813; Drug: Matching Placebo
- Part 2: JNJ-40411813 (Experimental): Participants will receive a single oral dose of JNJ-40411813 in Cohort 4.
  Interventions: Drug: JNJ-40411813
- Part 3: JNJ-40411813 or Matching Placebo (Experimental): Participants will receive a multiple oral dose of JNJ-40411813 or a matching placebo in Cohort 5 and optional Cohort 6.
  Interventions: Drug: JNJ-40411813; Drug: Matching Placebo

INTERVENTIONS:
Drug: JNJ-40411813 — JNJ-40411813 will be administered orally.
Drug: Matching Placebo — Matching placebo will be administered orally.
  Arms: Part 1: JNJ-40411813 or Matching Placebo; Part 3: JNJ-40411813 or Matching Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) after single dose and multiple dose administrations of JNJ-40411813 in Japanese healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* Be a Japanese man
* Be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Blood pressure (after the participant supine for 5 minutes) between 90 and 140 millimeter of Mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study intervention, a participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person. Male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak. Recommended highly effective methods of contraception in this study for female partners of male participants to use in addition to the male participant wearing a condom during include: a) oral hormonal contraception, b) intrauterine device, c) intrauterine hormone-releasing system, and d) bilateral tubal occlusion
* A participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum 90 days after receiving the last dose of study intervention

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at screening as deemed appropriate by the investigator
* Known allergies, hypersensitivity, or intolerance to JNJ-40411813 or its excipients
* Test positive for human immunodeficiency virus (HIV) antigen/antibodies, hepatitis A antibody immunoglobulin M (IgM), syphilis, hepatitis B surface antigen (HbsAg) or hepatitis C virus (HCV) antibodies at screening

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Parts 1 and 2: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 6 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Part 3: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 8 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Parts 1 and 2: Plasma Concentration of JNJ-40411813 | Predose, up to 96 hours postdose (Day 5)
  Plasma samples will be analyzed to determine concentrations of JNJ-40411813 using a validated, specific, and sensitive liquid chromatography mass spectrometry/mass spectrometry (LC-MS/MS).
Part 3: Plasma Concentration of JNJ-40411813 | Predose, up to 312 hours postdose (Day 14)
  Plasma samples will be analyzed to determine concentrations of JNJ-40411813 using a validated, specific, and sensitive LC-MS/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Souseikai Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinicaltrials/ transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency